CLINICAL TRIAL: NCT05576818
Title: Clinical Study Evaluating the Efficacy and Safety of Synbiotic as an Adjuvant Therapy in the Treatment of Parkinson's Disease
Brief Title: Effect of Synbiotic as an Adjuvant Therapy in the Treatment of Parkinson's Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ehab Sayed Ramadan, Demonstrator at clinical pharmacy department, faculty of pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Synbiotics Parkinson's disease
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Synbiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): this group will include 33 patients who will receive their standard dopamine replacement therapy for 3 months
- Synbiotic group (Active Comparator): this group will involve 33 patients who will receive Synbiotic preparation containing Lactobacillus acidophilus 10 billion colony forming unit (CFU) and prebiotic fibers 2 sachets daily together with their standard dopamine replacement therapy for 3 months
  Interventions: Drug: Lactobacillus acidophilus 10 billion colony forming unit (CFU) and prebiotic fibers

INTERVENTIONS:
Drug: Lactobacillus acidophilus 10 billion colony forming unit (CFU) and prebiotic fibers — Two sachets daily of synbiotic preparation containing Lactobacillus acidophilus 10 billion colony forming unit (CFU) and prebiotic fibers
  Other Names: Synbiotic
  Arms: Synbiotic group

SUMMARY:
This study aims to investigate the possible efficacy and safety of synbiotic preparation of Lactobacillus acidophilus probiotic with prebiotic fibers as an adjuvant therapy in the treatment of Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 65 years old
* Both sexes
* Patients with Parkinson's disease on dopamine replacement therapy
* Modified Hoehn and Yahr stage, MHY 1-4

Exclusion Criteria:

* Patients who are currently using or used antibiotics therapy in the preceding month
* Patients who are currently using or used other probiotic products in the preceding two weeks
* Patients scheduled to undergo GIT surgery or those underwent GIT surgery
* Patients with Known allergy to probiotics
* Patients receiving artificial enteral or intravenous nutrition
* Patients with depression and/or psychosis
* Patients taking antioxidant and/or anti-inflammatory medications
* Patients with Hyperthyroidism
* Patients with inflammatory condition and/or condition involving oxidative stress
* Smokers
* Modified Hoehn & Yahr stage MHY 5

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The change in MDS-Unified Parkinson's Disease Rating Scale. | 3 months
  Patients will undergo clinical assessment according to MDS-Unified Parkinson's Disease Rating Scale at baseline and after 3 months

SECONDARY OUTCOMES:
The change in the serum level of α-Synuclein | 3 months
  Blood samples will be collected at baseline and after 3 months
The change in the serum level of Tumor necrosis factor α (TNF α ) | 3 months
  Blood samples will be collected at baseline and after 3 months
The change in the serum level of Brain derived neurotrophic factor ( BDNF) | 3 months
  Blood samples will be collected at baseline and after 3 months
The change in the serum level of Malondialdehyde (MDA) | 3 months
  Blood samples will be collected at baseline and after 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramadan ME, Mostafa TM, Ghali AA, El-Afify DR. Randomized controlled trial evaluating synbiotic supplementation as an adjuvant therapy in the treatment of Parkinson's disease. Inflammopharmacology. 2025 Jul;33(7):3897-3908. doi: 10.1007/s10787-025-01752-8. Epub 2025 May 28. PMID 40434674